CLINICAL TRIAL: NCT01903928
Title: An Open Phase 2 Trial to Evaluate Safety of a Therapeutic Vaccine, ASP0113, in Recipients Undergoing Allogeneic Hematopoietic Cell Transplant (HCT)
Brief Title: A Study to Evaluate Safety and Tolerability of a Therapeutic Vaccine, ASP0113, in Subjects Undergoing Allogeneic Hematopoietic Cell Transplant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0113-CL-1003
Record Dates: First submitted 2013-07-01; First posted 2013-07-19 (Estimated); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Allogeneic Hematopoietic Cell Transplant
Keywords: cytomegalovirus; HCT; DNA vaccine; transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ASP0113 group (Experimental): Participants receive 1 mL of ASP0113 intramuscularly 5 times, on days -14 to -3, 14 to 40, 60 ± 5, 90 ± 10, and 180 ± 10, counting from the transplantation (stem cell transfusion) day (day 0)
  Interventions: Biological: ASP0113

INTERVENTIONS:
Biological: ASP0113 — injection

SUMMARY:
This study is to evaluate safety and tolerability of a therapeutic vaccine, ASP0113, in subjects undergoing allogeneic HCT. The occurrence of CMV viremia and immunogenicity are also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Subject is planned to undergo either of the following:

  * Sibling Donor Transplant - 7/8 Human Leukocyte Antigen (HLA)-A, -B, -C, -DRß1 match utilizing high resolution typing or 8/8 (HLA)-A, -B, -C, -DRß1 match utilizing low or high resolution typing.
  * Unrelated Donor Transplant - 7/8 or 8/8 HLA-A, -B, -C, -DRß1 match utilizing high resolution typing.
* Subject has one of the following underlying diseases: Acute myeloid leukemia (AML) /Acute lymphoblastic leukemia (ALL) / Acute undifferentiated leukemia (AUL) /Acute biphenotypic leukemia / Chronic myelogenous leukemia (CML) / Chronic lymphocytic leukemia (CLL) / myelodysplastic syndrome(s) (MDS)
* Subject is scheduled to receive an allogeneic peripheral blood stem cell (PBSC) or bone marrow transplant (BMT) for the treatment of hematologic disorders

Exclusion Criteria:

* Subject has active CMV disease or infection or has received treatment for active CMV disease or infection within 90 days prior to transplant
* Subject has planned CMV prophylactic therapy with antiviral drugs or CMV-specific immunoglobulins
* Subject has a modified hematopoietic cell transplant comorbidity index (HCT-CI) score > 3
* Subject is known to be positive for human immunodeficiency virus (HIV), hepatitis B surface antigen or hepatitis C ribonucleic acid (RNA)
* Subject has received any of the following substances or treatments:

  * T-cell depletion of donor cell product.
  * Alemtuzumab within 60 days prior to transplant, including conditioning regimen. Subjects for whom treatment with alemtuzumab is planned at any time from 60 days prior to through one year post-transplant should not be enrolled in the trial.
  * Administration of a CMV vaccine, including any prior exposure to ASP0113.
* Subject has received an allogeneic stem cell transplant within one year prior to transplant
* Subject has a current malignancy in addition to the malignancy being treated for the study or the subject has a history of any other malignancy
* Subject has an unstable medical or psychiatric condition, including a history of illicit drug(s) or alcohol abuse that the Investigator believes will interfere with protocol requirements.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2013-06-20 (Actual); Primary Completion 2015-01-19 (Actual); Study Completion 2015-01-19 (Actual)

PRIMARY OUTCOMES:
Safety assessed by the incidence of adverse events, vital signs, physical exam and labo-tests | for 365 days after HCT

SECONDARY OUTCOMES:
Local reactogenicity | for 14 days following each injection
  protocol-specified reactogenicity scale
Incidence of CMV viremia | for 365 days after HCT
  CMV plasma viral load ≥ 1000 copies
CMV-specified antiviral therapy | for 365 days after HCT
  CMV-specific AVT(Anti-virus therapy) initiated for a CMV plasma viral load ≥ 1000 copies
Incidence of cytomegalovirus end-organ disease (CMV EOD) | for 365 days after HCT
  CMV pneumonia, CMV gastroenteritis, CMV hepatitis, et al
Maximum grade of Graft Versus Host Disease (GVHD) | for 365 days after HCT

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (2):
- Japan (2):
  - Kantou
  - Kyushu

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Mori T, Kanda Y, Takenaka K, Okamoto S, Kato J, Kanda J, Yoshimoto G, Gondo H, Doi S, Inaba M, Kodera Y. Safety of ASP0113, a cytomegalovirus DNA vaccine, in recipients undergoing allogeneic hematopoietic cell transplantation: an open-label phase 2 trial. Int J Hematol. 2017 Feb;105(2):206-212. doi: 10.1007/s12185-016-2110-3. Epub 2016 Oct 28. PMID 27796740
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=285